CLINICAL TRIAL: NCT00885755
Title: A Prospective Study to Evaluate Alterations in Molecular Biomarkers in HER2 Neu Positive Metastatic Breast Cancer Together With Assessment of Trastuzumab Use Beyond Progression After Initial Response to Trastuzumab-taxane Based Treatment
Brief Title: A Study of Herceptin (Trastuzumab)and Biomarkers in Patients With HER2-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO22004; 2008-004013-94
Record Dates: First submitted 2009-03-16; First posted 2009-04-22 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Trastuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Standard taxane therapy; Drug: capecitabine [Xeloda]; Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: Standard taxane therapy — As prescribed
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid on days 1-14 of each 3-week cycle (only in patients who have progressed)
Drug: trastuzumab [Herceptin] — 8mg/kg iv loading dose on day 1 of first 3-week cycle, and 6mg/kg iv on day 1 of each subsequent cycle

SUMMARY:
This single arm study will evaluate alterations in molecular marker expression in HER2-positive targeted therapy, and will evaluate the effect of continued treatment with Herceptin and Xeloda beyond progression following initial Herceptin-taxane chemotherapy. Patients who develop progressive disease will receive first-line Herceptin (8mg/kg iv loading dose and 6mg/kg iv every 3 weeks) + taxane therapy. patients who develop progressive disease within 9 weeks of treatment will continue treatment with Herceptin in combination with Xeloda (1000mg/m2 po bid on days 1-14 of each 3-week cycle).Biopsies of tumor tissue will be taken for biomarker and gene profiling evaluation. The anticipated time on study treatment is until disease progression, intolerable side effects or patient choice, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* HER2-positive breast cancer;
* al least one metastatic site amenable for core biopsy;
* left ventricular ejection fraction >50%.

Exclusion Criteria:

* prior adjuvant/neoadjuvant Herceptin within past 6 months;
* prior adjuvant taxane therapy within past 12 months;
* use of chemotherapy, immunotherapy or biological anticancer therapy within past 3 weeks;
* known bleeding diatheses.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-08-13 (Actual); Primary Completion 2013-02-18 (Actual); Study Completion 2013-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Australia (6):
  - Royal Prince Alfred Hospital; Medical Oncology, Camperdown, New South Wales
  - Royal North Shore Hospital; Oncology, St Leonards, New South Wales
  - Eastern Health Breast Cancer Research, East Ringwood, Victoria
  - Border Medical Oncology; Murray Valley Private Hospital, Wodonga, Victoria
  - Mount Medical Center, Perth, Western Australia
  - Royal Perth Hospital; Department of Medical Oncology, Perth, Western Australia
- Spain (2):
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Sweden (2):
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- United Kingdom (3):
  - Hull Royal Infirmary, Hull
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Nottingham City Hospital; Oncology, Nottingham

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A:Trastuzumab+Taxane /Capecitabine (6 Weeks): This group included participants who progressed after at least six weeks of trastuzumab/taxane treatment. In Part I of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 milligrams per square meter (mg/m^2) or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. In Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on Body Surface Area (BSA) on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
- Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks: This group included participants who progressed within less than six weeks of trastuzumab/taxane treatment. In Part 1 of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. In Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on BSA on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
- No Group: This group included participants who died before any study disease assessments or post-baseline biopsies. In Part I of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression.
Period: Part I: Trastuzumab+Taxane
Arm/Group | Group A:Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks | No Group
Started | 31 | 1 | 1
Completed | 13 | 1 | 0
Not Completed | 18 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Unknown Reason | 16 | 0 | 0
Not completed — Sufficient Response Achieved | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1
Period: Part II: Trastuzumab + Capecitabine.
Arm/Group | Group A:Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks | No Group
Started | 13 | 1 | 0
Completed | 8 | 1 | 0
Not Completed | 5 | 0 | 0
Not completed — Unknown Reason | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All registered participants were included in the ITT population.
Groups:
- Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks): This group included participants who progressed after at least six weeks of trastuzumab/taxane treatment. In Part I of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. In Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on BSA on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
- Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks: This group included participants who progressed within less than six weeks of trastuzumab/taxane treatment. In Part I of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. In Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on BSA on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
- No Group: This group included participants who died before any on study disease assessments or post-baseline biopsies. In Part 1 of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression.
- Total: Total of all reporting groups
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks | No Group | Total
Number analyzed (Participants) | 31 | 1 | 1 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.73) | 37.0 (NA) — Standard deviation was not available since there was only 1 participant. | 85.0 (NA) — Standard deviation was not available since there was only 1 participant. | 55.9 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 1 | 1 | 33
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part I: Progression Free Survival (PFS) by Biomarker
Description: Progression was defined as an increase by at least 20 percent (%) from the smallest value in the Sum of Longest Diameter (SLD) of lesions. Biomarkers investigated: p95 human epidermal growth factor receptor 2 (p95HER2) positive (+ve) and negative (-ve) , insulin growth factor-1 receptor (IGF1R) less than (<) median and greater than or equal to (≥) median membrane H score, c-MET <median and ≥median membrane H score, phosphatase and tensin homolog gene (PTEN) <median and ≥median cytoplasm H score, HER2 <median and ≥median membrane H score, phosphatidylinositol-3-kinase (PI3K) catalytic subunit wild type (WT) and mutation (M), and FC gamma receptors IIIa homozygous Phenyl alanine (FF), heterozygous Phenyl alanine/Valine (VF) and homozygous Valine (VV), receptor IIa Phenotypes homozygous Histidine (HH), heterozygous Histidine/Arginine (HR) and homozygous Arginine (RR) IIb phenotypes homozygous Isoleucien (II),heterozygous Isoleucine/Threonine (IT) and homozygous Threonine (TT) .
Time Frame: End of first 2 Cycles (Weeks 3 and 6), every 3 Cycles for 18 weeks, then every 4 cycles until progression, unacceptable toxicity or participant decision to cease treatment up to 46 months
Population: Per Protocol (PP) population included all participants who had received a complete first dose of study medication and had baseline and at least one on-treatment biomarker assessment. Number (n) equals (=) number of participants with biomarker data available for the specified biomarker.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks): This group included participants who progressed after at least six weeks of trastuzumab/taxane treatment. In Part 1 of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. in Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on BSA on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 27 | 1
months
  p95 HER2 +ve (n=9,0) | NA [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  p95 HER2 -ve (n=15,1) | 13.963 [7.261 to 22.407] | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  IGF1R <median (n=12,0) | 12.649 [4.698 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  IGF1R ≥median (n=14,1) | 22.209 [7.261 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET <median (n=10,1) | 18.595 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET ≥median (n=15,0) | 13.733 [7.031 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN <median (n=12,0) | 22.209 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN ≥median (n=14,1) | 13.963 [6.374 to 31.179] | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 <median (n=11,1) | 13.733 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 ≥median (n=14,0) | 22.209 [7.031 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PI3K Amino Acids WT (n=17,1) | 13.848 [7.261 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  PI3K Amino Acids M (n=9,0) | 22.407 [4.698 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V FF (n=9,0) | 10.612 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V VF (n=5,1) | 11.335 [9.528 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIIa F176V VV (n=4,0) | 22.407 [22.209 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH (n=3,0) | NA [9.528 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HR (n=8,1) | 22.209 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIa R166H RR (n=8,0) | 13.963 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T II (n=12,1) | 11.335 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIb I232T IT (n=1,0) | NA [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T TT (n=1,0) | NA [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
Statistical Analysis 1: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Positive / Negative) for the biomarker p95; Test type: Superiority or Other; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.109 to 1.535]
Statistical Analysis 2: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression: Hazard ratio (Membrane H-Score: <median / ≥median) for the biomarker IGF1R; Test type: Superiority or Other; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.430 to 3.282]
Statistical Analysis 3: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Membrane H-Score: <median / ≥median) for the biomarker c-MET; Test type: Superiority or Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.306 to 2.425]
Statistical Analysis 4: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Cytoplasm H-Score: <median / ≥median) for the biomarker PTEN; Test type: Superiority or Other; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.164 to 1.453]
Statistical Analysis 5: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Membrane H-Score: < median / ≥median) for the biomarker HER2; Test type: Superiority or Other; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.377 to 3.160]
Statistical Analysis 6: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Mutation Status: Wild type / Mutation) for the biomarker PI3K amino acids; Test type: Superiority or Other; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.409 to 4.132]
Statistical Analysis 7: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: FF / VF) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.183, 95% CI 2-sided [0.226 to 6.197]
Statistical Analysis 8: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: FF / VV) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.989, 95% CI 2-sided [0.378 to 10.470]
Statistical Analysis 9: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: VF / VV) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.732, 95% CI 2-sided [0.235 to 12.783]
Statistical Analysis 10: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: HH / HR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Hazard Ratio (HR) = 0.576, 95% CI 2-sided [0.067 to 4.968]
Statistical Analysis 11: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: HH / RR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Hazard Ratio (HR) = 0.743, 95% CI 2-sided [0.082 to 6.720]
Statistical Analysis 12: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: HR / RR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.274 to 4.199]

2. Secondary Outcome: Part I: TTP in Intent to Treat (ITT) Population
Description: TTP was determined as the time in months from the date of screening until first progression. In participants with measurable disease, progression was defined according to RECIST (SLD increased by at least 20% from the smallest value on study [including baseline, if that is the smallest]). In participants with non-measurable disease, progression was defined as the presence of new lesions or unequivocal progression during treatment.
Time Frame: as for outcome 1
Population: ITT population; Participant from Group B and from No group were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 31 | 1
months | 22.21 [9.53 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.22 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.

3. Primary Outcome: Part II: Progression Free Survival (PFS) by Biomarker
Description: PFS was calculated from first study medication in Part II to date of progression or death.The relationship between PFS and the following biomarker variables was investigated in each of study Part 1 and 2: p95HER2 +ve and -ve population, IGF1R <median and ≥ median membrane H score, c-MET <median and ≥median membrane H score, PTEN <median and ≥median cytoplasm H score, HER2 <median and ≥median membrane H score, PI3K catalytic subunit WT and M, and FC gamma receptors IIIa, IIa and IIb Phenotypes FF, VF and VV, HH, HR and RR, and II, IT and TT.
Time Frame: as for outcome 1
Population: PP population; n = number of participants with biomarker data available for the specified biomarker.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 27 | 1
months
  p95 +ve (n=2,0) | 8.148 [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  p95 -ve (n=5,1) | 3.450 [0.854 to 8.115] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  IGF1R <median (n=4,0) | 8.115 [0.854 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  IGF1R ≥median (n=4,1) | 4.074 [1.971 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET<median (n=3,1) | 4.698 [3.450 to 4.698] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET≥median (n=4,0) | 5.043 [0.854 to 8.148] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN <median (n=4,0) | 4.698 [1.971 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN ≥median (n=3,1) | 3.450 [0.854 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 <median (n=2,1) | 8.148 [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 ≥median (n=5,0) | 3.450 [0.854 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PI3K Amino Acids WT (n=10,1) | 5.651 [1.971 to 24.214] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  PI3K Amino Acids M (n=2,0) | 4.485 [0.854 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V FF (n=4,0) | 4.320 [0.854 to 8.148] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V VF (n=2,1) | 13.832 [3.450 to 24.214] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIIa F176V VV (n=2,0) | NA [NA to NA] — Data are not available since there was no evaluable participant. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH (n=1,0) | 3.450 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HR (n=5,1) | 8.115 [0.854 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIa R166H RR (n=3,0) | 5.651 [2.990 to 24.214] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T II (n=7,1) | 5.651 [0.854 to 24.214] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.

4. Primary Outcome: Part I: Time to Progression (TTP) by Biomarker
Description: Progression was defined as an increase by at least 20% from the smallest value in the SLD of lesions.TTP was determined as the time in months from the date of screening until first progression.The relationship between PFS and the following biomarker variables was investigated in each of study Part 1 and 2: p95 HER2 +ve and -ve population, IGF1R <median and ≥median, c-MET <median and ≥median, PTEN <median and ≥median, HER2 <median and ≥median, PI3K catalytic subunit WT and M, and FC gamma receptors IIIa, IIa and IIb Phenotypes FF, VF and VV, HH, HR and RR, and II, IT and TT . The correlation between the biomarker variables and TTP were investigated using a univariate Cox regression model and time-to-event methods (Kaplan-Meier).
Time Frame: End of first 2 Cycles (Weeks 3 and 6), every 3 Cycles for 18 weeks, then every 4 cycles until progression, unacceptable toxicity or participant decision to cease treatment up to 46 weeks
Population: PP population; n = number of participants with biomarker data available for the specified biomarker.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 27 | 1
months
  p95 +ve (n=9,0) | NA [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  p95 -ve (n=15,1) | 13.963 [7.261 to 22.407] | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  IGF1R <median (n=12,0) | 11.335 [4.698 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  IGF1R ≥median (n=14,1) | 22.407 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET <median (n=10,1) | 31.179 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET ≥median (n=15,0) | 22.209 [6.374 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  PTEN <median (n=12,0) | 22.209 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN ≥median (n=14,1) | 13.963 [6.374 to 31.179] | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 <median (n=11,1) | NA [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 ≥median (n=14,0) | 22.209 [7.031 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PI3K Amino Acids WT (n=17,1) | 13.963 [7.261 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  PI3K Amino Acids M (n=9,00) | 22.407 [4.698 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V FF (n=9,0) | 13.963 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V VF (n=5,1) | 11.335 [9.528 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIIa F176V VV (n=4,0) | 22.407 [22.209 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH (n=3,0) | NA [9.528 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HR (n=8,1) | 22.209 [3.384 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIa R166H RR (n=8,0) | 13.963 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T II (n=12,1) | 13.963 [5.914 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.216 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIb I232T IT (n=1,0) | NA [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T TT (n=1,0) | NA [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
Statistical Analysis 1: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Positive / Negative) for the biomarker p95 HER2; Test type: Superiority or Other; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.120 to 1.790]
Statistical Analysis 2: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regressionHazard ratio (Membrane H-Score: <median / ≥median) for the biomarker IGF1R; Test type: Superiority or Other; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.394 to 3.518]
Statistical Analysis 3: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Membrane H-Score: < median / ≥median) for the biomarker c-met; Test type: Superiority or Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.268 to 2.514]
Statistical Analysis 4: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Cytoplasm H-Score: < median / ≥median) for the marker PTEN; Test type: Superiority or Other; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.183 to 1.768]
Statistical Analysis 5: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Membrane H-Score: < median / ≥median) for the biomarker HER2; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.242 to 2.733]
Statistical Analysis 6: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regressionHazard ratio (Mutation Status: Wild type / Mutation) for the biomarker PI3K amino acids; Test type: Superiority or Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.337 to 3.632]
Statistical Analysis 7: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Hazard ratio (Phenotype: FF / VF) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Hazard Ratio (HR) = 0.957, 95% CI 2-sided [0.172 to 5.336]
Statistical Analysis 8: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Hazard ratio (Phenotype: FF / VV) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.666, 95% CI 2-sided [0.298 to 9.305]
Statistical Analysis 9: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Hazard ratio (Phenotype: VF / VV) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.732, 95% CI 2-sided [0.235 to 12.783]
Statistical Analysis 10: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: HH / HR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Hazard Ratio (HR) = 0.576, 95% CI 2-sided [0.067 to 4.968]
Statistical Analysis 11: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: HH / RR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Hazard Ratio (HR) = 0.956, 95% CI 2-sided [0.098 to 9.319]
Statistical Analysis 12: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate Cox regression Hazard ratio (Phenotype: HR / RR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Hazard Ratio (HR) = 1.292, 95% CI 2-sided [0.296 to 5.640]

5. Secondary Outcome: Part I: PFS in ITT Population
Description: PFS was determined as the time in months from the date of screening until first progression. In participants with measurable disease, progression was defined according to RECIST (SLD increased by at least 20% from the smallest value on study [including baseline, if that is the smallest]).. In participants with non-measurable disease, progression was defined as the presence of new lesions or unequivocal progression during treatment.
Time Frame: as for outcome 1
Population: ITT population; Participant from Group B and from No group were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 31 | 1
months | 18.60 [8.08 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 1.22 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.

6. Secondary Outcome: Part II: TTP in Intent to Treat (ITT) Population
Description: TTP was calculated from first study medication in Part II to date of progression. In participants with measurable disease progression was defined according to RECIST(SLD increased by at least 20% from the smallest value on study [including baseline, if that is the smallest]). In participants with non-measurable disease, progression was defined as the presence of new lesions or unequivocal progression during treatment.
Time Frame: as for outcome 1
Population: ITT population; Participant from Group B and from No group were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 13 | 1
months | 5.65 [2.99 to 8.15] | 13.83 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.

7. Secondary Outcome: Part II: PFS in ITT Population
Description: PFS was calculated from first study medication in Part II to date of progression or death. In participants with measurable disease progression was defined according to RECIST (SLD increased by at least 20% from the smallest value on study [including baseline, if that is the smallest]). In participants with non-measurable disease, progression was defined as the presence of new lesions or unequivocal progression during treatment.
Time Frame: as for outcome 1
Population: ITT population; Participant from Group B and from No group were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 13 | 1
months | 5.65 [2.99 to 24.21] | 13.83 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.

8. Secondary Outcome: Overall Survival in Per Protocol Population
Description: Overall survival was calculated in months from the day of screening until death.
Time Frame: End of first 2 Cycles (Weeks 3 and 6), every 3 cycles for 18 weeks, then every 4 cycles until death (up to 46 months)
Population: PP population
Measure: Median (Full Range); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks)
Number analyzed (Participants) | 27
months | 36.40 [6.57 to 40.28]

9. Secondary Outcome: Overall Survival in ITT Population
Description: Overall survival was calculated in months from the day of screening until death.
Time Frame: End of first 2 Cycles (Weeks 3 and 6), every 3 cycles for 18 weeks, then every 4 cycles until death (up to 46 months)
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks)
Number analyzed (Participants) | 31
months | NA [6.57 to 40.28] — Estimate Not Available due to insufficient follow-up to allow estimation.

10. Secondary Outcome: Part I and II: Percentage of Participants With a Best Overall Response of CR or PR in ITT Population
Description: Best Overall response was defined according to RECIST. CR: disappearance of all target lesions and all pathological lymph nodes below 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions.
Time Frame: as for outcome 1
Population: ITT population; n = number of participants analyzed for the specified category.
Measure: Number; unit: percentage of participants
Groups:
- Group A: Trastuzumab+Taxane /Capcetabine (6 Weeks): This group included participants who progressed after at least six weeks of trastuzumab/taxane treatment. In Part I of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. In Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on BSA on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
Arm/Group | Group A: Trastuzumab+Taxane /Capcetabine (6 Weeks)
Number analyzed (Participants) | 20
percentage of participants
  Part I: Responders (n=20) | 75.0
  Part I: Non-Responders (n=20) | 20.0
  Part I: Missing (n=20) | 5.0
  Part II: Responders (n=9) | 11.1
  Part II: Non-Responders (n=9) | 88.9
  Part II: Missing (n=9) | 0.0

11. Primary Outcome: Part II: TTP by Biomarker
Description: TTP was calculated from first study medication in Part II to date of progression. The relationship between TTP and the following biomarker variables was investigated in each of study Part 1 and 2: p95 HER2 +ve and -ve population, IGF1R <median and ≥median, c-MET <median and ≥median, PTEN <median and ≥median, HER2 <median and ≥median, PI3K catalytic subunit WT and M, and FC gamma receptors IIIa, IIa and IIb Phenotypes FF, VF and VV, HH, HR and RR, and II, IT and TT .
Time Frame: as for outcome 1
Population: PP population; n = number of participants with biomarker data available for the specified biomarker.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks) | Group B: Trastuzumab+Taxane/ Capecitabine <6 Weeks
Number analyzed (Participants) | 27 | 1
months
  p95 HER2 +ve (n=2,0) | 8.148 [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  p95 HER2 -ve (n=5,1) | 3.450 [0.854 to 8.115] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  IGF1R <median (n=4,0) | 8.115 [0.854 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  IGF1R ≥median (n=4,1) | 4.074 [1.971 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET <median (n=3,1) | 4.698 [3.450 to 4.698] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  c-MET ≥median (n=4,0) | 5.043 [0.854 to 8.148] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN <median (n=4,0) | 4.698 [1.971 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PTEN ≥median (n=3,1) | 3.450 [0.854 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 <median (n=2,1) | 8.148 [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  HER2 ≥median (n=5,0) | 3.450 [0.854 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  PI3K Amino Acids WT (n=10,1) | 5.651 [1.971 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  PI3K Amino Acids M (n=2,0) | 4.485 [0.854 to 8.115] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V FF (n=4,0) | 4.320 [0.854 to 8.148] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIIa F176V VF (n=2,1) | NA [3.450 to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIIa F176V VV (n=2,0) | NA [NA to NA] — Data are not available since there was no evaluable participant. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH (n=1,0) | 3.450 [NA to NA] — Estimate Not Available due to insufficient follow-up to allow estimation. | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HR (n=5,1) | 8.115 [0.854 to 8.148] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.
  FC Gamma Receptor IIa R166H RR (n=3,0) | 5.651 [2.990 to 5.651] | NA [NA to NA] — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T II (n=7,1) | 5.651 [0.854 to 8.115] | 13.832 [NA to NA] — Confidence Interval was not applicable since there was only 1 participant.

12. Primary Outcome: Part I: Percentage of Participants With a Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progrerssive Disease (PD) by Biomarker
Description: BOR was defined according to the Response Evaluation Criteria In Solid Tumors (RECIST). CR: disappearance of all target lesions and all pathological lymph nodes below 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions. The relationship between best response and the following biomarkers was investigated: p95 HER2 (+ve/-ve), IGF1R, c-MET, PTEN, HER2 (median/≥median), PI3K catalytic subunit (WT/M), and FC gamma receptors IIIa, IIa and IIb (phenotypes FF, VF, VV, HH, HR, RR and II, IT and TT respectively). The correlation between the biomarker variables and percentage of participants with best response were investigated using a univariate regression analysis.
Time Frame: as for outcome 4
Population: PP population; n = number of participants with biomarker data available for the specified biomarker. Data are reported for Group A only as there were no evaluable participants in Group B.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks)
Number analyzed (Participants) | 19
percentage of participants
  p95 HER2 +ve CR (n=5) | 0.0
  p95 HER2 +ve PR (n=5) | 25.0
  p95 HER2 +ve SD (n=5) | 50.0
  p95 HER2 +ve PD (n=5) | 25.0
  p95 HER2 -ve CR (n=12) | 0.0
  p95 HER2 -ve PR (n=12) | 91.7
  p95 HER2 -ve SD (n=12) | 8.3
  p95 HER2 -ve PD (n=12) | 0.0
  IGF1R < median CR (n=9) | 0.0
  IGF1R < median PR (n=9) | 62.5
  IGF1R < median SD (n=9) | 37.5
  IGF1R < median PD (n=9) | 0.0
  IGF1R ≥median CR (n=9) | 0.0
  IGF1R ≥median PR (n=9,0) | 88.9
  IGF1R ≥median SD (n=9) | 0.0
  IGF1R ≥median PD (n=9) | 11.1
  c-MET <median CR (n=6) | 0.0
  c-METt <median PR (n=6) | 83.3
  c-MET <median SD (n=6) | 0.0
  c-MET <median PD (n=6) | 16.7
  c-MET ≥median CR (n=11) | 0.0
  c-MET ≥median PR (n=11) | 70.0
  c-MET ≥median SD (n=11) | 30.0
  c-MET ≥median PD (n=11) | 0.0
  PTEN <median CR (n=6) | 0.0
  PTEN <median PR (n=6) | 83.3
  PTEN <median SD (n=6) | 16.7
  PTEN <median PD (n=6) | 0.0
  PTEN ≥median CR (n=12) | 0.0
  PTEN ≥median PR (n=12) | 72.7
  PTEN ≥median SD (n=12) | 18.2
  PTEN ≥median PD (n=12) | 9.1
  HER2 <median CR (n=8) | 0.0
  HER2 <median PR (n=8) | 75.0
  HER2 <median SD (n=8) | 12.5
  HER2 <median PD (n=8) | 12.5
  HER2 ≥median CR (n=10) | 0.0
  HER2 ≥median PR (n=10) | 77.8
  HER2 ≥median SD (n=10) | 22.2
  HER2 ≥median PD (n=10) | 0.0
  PI3K Amino Acids WT CR (n=11) | 0.0
  PI3K Amino Acids WT PR (n=11,0) | 90.0
  PI3K Amino Acids WT SD (n=11) | 0.0
  PI3K Amino Acids WT PD (n=11) | 10.0
  PI3K Amino Acids M CR (n=7) | 0.0
  PI3K Amino Acids M PR (n=7,0) | 57.1
  PI3K Amino Acids M SD (n=7) | 42.9
  PI3K Amino Acids M PD (n=7) | 0.0
  FC Gamma Receptor IIIa F176V FF CR (n=6) | 16.7
  FC Gamma Receptor IIIa F176V FF PR (n=6) | 50.0
  FC Gamma Receptor IIIa F176V FF SD (n=6) | 16.7
  FC Gamma Receptor IIIa F176V FF PD (n=6) | 16.7
  FC Gamma Receptor IIIa F176V VF CR (n=4) | 0.0
  FC Gamma Receptor IIIa F176V VF PR (n=4) | 66.7
  FC Gamma Receptor IIIa F176V VF SD (n=4) | 33.3
  FC Gamma Receptor IIIa F176V VF PD (n=4) | 0.0
  FC Gamma Receptor IIIa F176V VV CR (n=2) | 0.0
  FC Gamma Receptor IIIa F176V VV PR (n=2) | 100.0
  FC Gamma Receptor IIIa F176V VV SD (n=2) | 0.0
  FC Gamma Receptor IIIa F176V VV PD (n=2) | 0.0
  FC Gamma Receptor IIa R166H HH CR (n=3) | 33.3
  FC Gamma Receptor IIa R166H HH PR (n=3) | 66.7
  FC Gamma Receptor IIa R166H HH SD (n=3) | 0.0
  FC Gamma Receptor IIa R166H HH PD (n=3) | 0.0
  FC Gamma Receptor IIa R166H HR CR (n=5) | 0.0
  FC Gamma Receptor IIa R166H HR PR (n=5) | 25.0
  FC Gamma Receptor IIa R166H HR SD (n=5) | 50.0
  FC Gamma Receptor IIa R166H HR PD (n=5) | 25.0
  FC Gamma Receptor IIa R166H RR CR (n=5) | 0.0
  FC Gamma Receptor IIa R166H RR PR (n=5) | 80.0
  FC Gamma Receptor IIa R166H SD RR (n=5) | 20.0
  FC Gamma Receptor IIa R166H RR PD (n=5) | 0.0
  FC Gamma Receptor IIb I232T II CR (n=8) | 12.5
  FC Gamma Receptor IIb I232T II PR (n=8) | 50.0
  FC Gamma Receptor IIb I232T II SD (n=8) | 37.5
  FC Gamma Receptor IIb I232T II PD (n=8) | 0.0
  FC Gamma Receptor IIb I232T IT CR (n=1) | 0.0
  FC Gamma Receptor IIb I232T IT PR (n=1) | 100.0
  FC Gamma Receptor IIb I232T IT SD (n=1) | 0.0
  FC Gamma Receptor IIb I232T IT PD (n=1) | 0.0
Statistical Analysis 1: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (Positive / Negative) for the biomarker p95 HER 2; Test type: Superiority or Other; Odds Ratio (OR) = 0.030, 95% CI 2-sided [0.001 to 0.641]
Statistical Analysis 2: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (Membrane H-Score: ≥median /<median) for the biomarker IGF1R; Test type: Superiority or Other; Odds Ratio (OR) = 0.208, 95% CI 2-sided [0.017 to 2.600]
Statistical Analysis 3: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (Membrane H-Score: ≥ median /<median) for the biomarker c-MET; Test type: Superiority or Other; Odds Ratio (OR) = 2.143, 95% CI 2-sided [0.169 to 27.103]
Statistical Analysis 4: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (Cytoplasm H-Score: ≥ median /< median) for the biomarker PTEN; Test type: Superiority or Other; Odds Ratio (OR) = 1.875, 95% CI 2-sided [0.150 to 23.396]
Statistical Analysis 5: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (Membrane H-Score: ≥median /< median) for the biomarker HER2; Test type: Superiority or Other; Odds Ratio (OR) = 0.857, 95% CI 2-sided [0.091 to 8.075]
Statistical Analysis 6: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (PI3K mutation status: WT versus M) for the biomarker PI3K Amino Acids; Test type: Superiority or Other; Odds Ratio (OR) = 0.148, 95% CI 2-sided [0.012 to 1.900]
Statistical Analysis 7: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regressionOdds ratio (Phenotype: FF / VF) for the biomarker FC Gamma Receptor IIIa F176V; Test type: Superiority or Other; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.053 to 18.915]
Statistical Analysis 8: Comparison: Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks); Univariate logistic regression Odds ratio (Phenotype: HR / RR) for the biomarker FC Gamma Receptor IIa R166H; Test type: Superiority or Other; Odds Ratio (OR) = 0.083, 95% CI 2-sided [0.004 to 1.945]

13. Primary Outcome: Part II: Percentage of Participants With a Best Overall Response of CR, PR, SD or PD by Biomarker
Description: Best Overall response was defined according to RECIST. CR: disappearance of all target lesions and all pathological lymph nodes below 10 mm.PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions. The relationship between best response and the following biomarkers was investigated: p95 HER2 (+ve/-ve), IGF1R, c-MET, PTEN, HER2 (<median/≥median) , PI3K catalytic subunit (WT/M), and FC gamma receptors IIIa, IIa and IIb (phenotypes FF, VF, VV, HH, HR, RR and II, IT and TT respectively). The correlation between the biomarker variables and percentage of participants with best response were investigated using a univariate regression analysis.
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks)
Number analyzed (Participants) | 19
percentage of participants
  p95 HER2 +ve CR (n=2) | 0.0
  p95 HER2 +ve PR (n=2) | 0.0
  p95 HER2 +ve SD (n=2) | 100.0
  p95 HER2 +ve PD (n=2) | 0.0
  p95 HER2 -ve CR (n=4) | 0.0
  p95 HER2 -ve PR (n=4) | 0.0
  p95 HER2 -ve SD (n=4) | 50.0
  p95 HER2 -ve PD (n=4) | 50.0
  IGF1R <median CR (n=3) | 0.0
  IGF1R <median PR (n=3) | 0.0
  IGF1R <median SD (n=3) | 66.7
  IGF1R <median PD (n=3) | 33.3
  IGF1R ≥median CR (n=3) | 0.0
  IGF1R ≥median PR (n=3) | 0.0
  IGF1R ≥median SD (n=3) | 66.7
  IGF1R ≥median PD (n=3) | 33.3
  c-MET <median CR (n=2) | 0.0
  c-MET <median PR (n=2) | 0.0
  c-MET <median SD (n=2) | 100.0
  c-MET <median PD (n=2) | 0.0
  c-MET ≥median CR (n=4) | 0.0
  c-MET ≥median PR (n=4) | 0.0
  c-MET ≥median SD (n=4) | 50.0
  c-MET ≥median PD (n=4) | 50.0
  PTEN <median CR (n=4) | 0.0
  PTEN <median PR (n=4) | 0.0
  PTEN <median SD (n=4) | 75.0
  PTEN <median PD (n=4) | 25.0
  PTEN ≥median CR (n=2) | 0.0
  PTEN ≥median PR (n=2) | 0.0
  PTEN ≥median SD (n=2) | 50.0
  PTEN ≥median PD (n=2) | 50.0
  HER2 <median CR (n=2) | 0.0
  HER2 <median PR (n=2) | 0.0
  HER2 <median SD (n=2) | 100.0
  HER2 <median PD (n=2) | 0.0
  HER2 ≥median CR (n=4) | 0.0
  HER2 ≥median PR (n=4) | 0.0
  HER2 ≥median SD (n=4) | 50.0
  HER2 ≥median PD (n=4) | 50.0
  PI3K Amino Acids WT CR (n=7) | 0.0
  PI3K Amino Acids WT PR (n=7) | 14.3
  PI3K Amino Acids WT SD (n=7) | 71.4
  PI3K Amino Acids WT PD (n=7) | 14.3
  PI3K Amino Acids M CR (n=2) | 0.0
  PI3K Amino Acids M PR (n=2) | 0.0
  PI3K Amino Acids M SD (n=2) | 50.0
  PI3K Amino Acids M PD (n=2) | 50.0
  FC Gamma Receptor IIIa F176V FF CR (n=3) | 0.0
  FC Gamma Receptor IIIa F176V FF PR (n=3) | 0.0
  FC Gamma Receptor IIIa F176V FF SD (n=3) | 66.7
  FC Gamma Receptor IIIa F176V FF PD (n=3) | 33.3
  FC Gamma Receptor IIIa F176V VF CR (n=1) | 0.0
  FC Gamma Receptor IIIa F176V VF PR (n=1) | 0.0
  FC Gamma Receptor IIIa F176V VF SD (n=1) | 100.0
  FC Gamma Receptor IIIa F176V VF PD (n=1) | 0.0
  FC Gamma Receptor IIIa F176V VV CR (n=1) | 0.0
  FC Gamma Receptor IIIa F176V VV PR (n=1) | 100.0
  FC Gamma Receptor IIIa F176V VV SD (n=1) | 0.0
  FC Gamma Receptor IIIa F176V VV PD (n=1) | 0.0
  FC Gamma Receptor IIa R166H HH CR (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH PR (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH SD (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HH PD (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIa R166H HR CR (n=5) | 0.0
  FC Gamma Receptor IIa R166H HR PR (n=4) | 25.0
  FC Gamma Receptor IIa R166H HR SD (n=4) | 50.0
  FC Gamma Receptor IIa R166H HR PD (n=4) | 25.0
  FC Gamma Receptor IIa R166H RR CR (n=4) | 0.0
  FC Gamma Receptor IIa R166H RR PR (n=2) | 0.0
  FC Gamma Receptor IIa R166H RR SD (n=2) | 100.0
  FC Gamma Receptor IIa R166H RR PD (n=2) | 0.0
  FC Gamma Receptor IIb I232T II CR (n=4) | 0.0
  FC Gamma Receptor IIb I232T II PR (n=4) | 0.0
  FC Gamma Receptor IIb I232T II SD (n=4) | 75.0
  FC Gamma Receptor IIb I232T II PD (n=4) | 25.0
  FC Gamma Receptor IIb I232T IT CR (N=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T IT PR (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T IT SD (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T IT PD (n=0) | NA — Data are not available since there was no evaluable participant.
  FC Gamma Receptor IIb I232T TT CR (n=4) | 0.0
  FC Gamma Receptor IIb I232T TT PR (n=4) | 0.0
  FC Gamma Receptor IIb I232T TT SD (n=4) | 75.0
  FC Gamma Receptor IIb I232T TT PD (n=4) | 25.0

14. Secondary Outcome: Part I and II: Percentage of Participants With a Response by Best Overall Response by CR, PR, SD or PD in ITT Population
Description: as for outcome 10
Time Frame: as for outcome 1
Population: ITT population; n = number of participants analyzed for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Trastuzumab+Taxane /Capecitabine (6 Weeks)
Number analyzed (Participants) | 20
percentage of participants
  Part I: CR (n=20) | 5.0
  Part I: PR (n=20) | 70.0
  Part I: SD (n=20) | 15.0
  Part I: PD (n=20) | 5.0
  Part I: Missing (n=20) | 5.0
  Part II: CR (n=9) | 0.0
  Part II: PR (n=9) | 11.1
  Part II: SD (n=9) | 66.7
  Part II: PD (n=9) | 22.2
  Part II: Missing (n=9) | 0.0

ADVERSE EVENTS:
Time Frame: From the date of Screening until 4 weeks after the last visit of the participant
Groups:
- All Participants: In Part 1 of the study, participants received standard first-line therapy with trastuzumab and, at the discretion of treating clinician, either paclitaxel or docetaxel. Trastuzumab was administered according to SMPC. Paclitaxel and docetaxel were administered according to one of following regimens: docetaxel 75 mg/m^2 or 100 mg/m^2 3-weekly (if docetaxel-naïve) or docetaxel 75 mg/m^2 3-weekly (if prior adjuvant docetaxel) or docetaxel 60 mg/m^2 3-weekly (if liver dysfunction due to metastatic involvement) or paclitaxel 80 mg/m^2 weekly or 175 mg/m^2 3-weekly until first disease progression. in Part II of the study, participants received capecitabine twice-daily 1000 mg/m^2 or higher, calculated based on BSA on days 1 to 14 while continuing trastuzumab treatment per standard practice until disease progression, unmanageable toxicity or participant request for discontinuation.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 9/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=33)
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Medical device complication (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=33)
Diarrhoea (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 21
Influenza like illness (General disorders) | 12
Oedema peripheral (General disorders) | 11
Asthenia (General disorders) | 6
Mucosal inflammation (General disorders) | 6
Pain (General disorders) | 7
Chest pain (General disorders) | 6
Oedema (General disorders) | 4
Axillary pain (General disorders) | 3
Chest discomfort (General disorders) | 3
Chills (General disorders) | 3
Pyrexia (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 22
Nail disorder (Skin and subcutaneous tissue disorders) | 23
Palmer-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 16
Scab (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Onycholsis (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 16
Dysgeusia (Nervous system disorders) | 10
Neuropathy peripheral (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 5
Neurotoxicity (Nervous system disorders) | 4
Polyneuropathy (Nervous system disorders) | 3
Cognitive disorder (Nervous system disorders) | 2
Sinus headache (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Restless leg syndrome (Nervous system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 7
Rhinitis (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 5
Nail infection (Infections and infestations) | 4
Localised infection (Infections and infestations) | 2
Nail bed infection (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Skin infection (Infections and infestations) | 3
Herpes simplex (Infections and infestations) | 2
Hordeolum (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Procedural pain (Injury, poisoning and procedural complications) | 11
Fall (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 3
Arthropod bite (Injury, poisoning and procedural complications) | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 2
Conjunctivitis (Eye disorders) | 5
Dry eye (Eye disorders) | 5
Lacrimation increased (Eye disorders) | 4
Ocular surface disease (Eye disorders) | 3
Vision blurred (Eye disorders) | 3
Eye pain (Eye disorders) | 2
Hot flush (Vascular disorders) | 9
Lymphoedema (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Insomnia (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 12
Breast pain (Reproductive system and breast disorders) | 5
Menstruation irregular (Reproductive system and breast disorders) | 3
Amenorrhoea (Reproductive system and breast disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Drug hypersensitivity (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 2
Haemoglobin decreased (Investigations) | 2
Ejection fraction decreased (Investigations) | 2
Weight increased (Investigations) | 2
Palpitations (Cardiac disorders) | 2
Left ventricular dysfunction (Cardiac disorders) | 2

LIMITATIONS AND CAVEATS:
The study was prematurely terminated on December 31, 2012. The end of study follow-up was February 18, 2013.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.